CLINICAL TRIAL: NCT05459285
Title: Pharmacokinetics, Safety and Immunogenicity of 14028 Injection Versus Dulaglutide Injection in Healthy Subjects: a Phase I ，Single-center, Randomized, Open-label, Single-dose, Parallel-controlled Clinical Study
Brief Title: A Pharmacokinetic Study Comparing the 14028 Injection and TRULICITY® in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14028-DM-101
Record Dates: First submitted 2022-07-08; First posted 2022-07-14 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 14028 injection (Experimental): Subjects receive 14028 injection in the study, 0.75mg, once
  Interventions: Biological: 14028 injection
- dulaglutide injection (TRULICITY®) (Active Comparator): Subjects receive dulaglutide injection (TRULICITY®) in the study, 0.75mg, once
  Interventions: Biological: dulaglutide injection

INTERVENTIONS:
Biological: 14028 injection — 14028 injection, single dose, s.c. injection
  Arms: 14028 injection
Biological: dulaglutide injection — dulaglutide injection(TRULICITY®), single dose, s.c. injection
  Other Names: TRULICITY®
  Arms: dulaglutide injection (TRULICITY®)

SUMMARY:
To evaluate the pharmacokinetics similarity between the 14028 injection produced by Sunshine Lake Pharma Co., Ltd. and dulaglutide injection (TRULICITY®) produced by Eli Lilly and Company for single dose in healthy male subjects, as well as to evaluate the similarity of the safety and immunogenicity between 14028 Injection and TRULICITY® in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the trial, understand and comply with the research process, and participate the trial voluntarily
2. Healthy male subjects aged 18 to 45 (including the critical value)
3. Weight > or = 50 kg, and 19.0 kg/m2 < or = BMI (body mass index) < or = 28.0 kg/m2
4. Vital signs, physical examination, laboratory examination, electrocardiogram, thyroid color Doppler ultrasound, abdominal color Doppler ultrasound and chest X-ray (anteroposterior) and other test results during screening are normal or have no clinical significance as judged by the investigator
5. Subjects agree to use effective contraceptive methods from signing the informed consent form to the end of the trial drug use within 3 months, and there is no sperm donation plan.

Exclusion Criteria:

1. The investigator judges that the subjects have the following clinically significant diseases (including but not limited to gastrointestinal, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases)
2. Have a medical or family history of medullary thyroid cancer (grandparents, parents, brothers and sisters), or a genetic disease that lead to medullary thyroid cancer; or a history or family history of multiple endocrine neoplasia syndrome type 2
3. Past or current history of pancreatitis (chronic or acute pancreatitis)
4. Past or current history of habitual constipation or intestinal obstruction
5. Clinically significant history of drug allergy or specific allergic disease (asthma, urticaria) or known allergy to the investigational drug and any component or related excipient components
6. Those who have difficulty with venous blood collection, a history of needle sickness, haemorrhage, or a known tendency to severe bleeding
7. Positive test results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), human immunodeficiency virus antibody (HIV), and Treponema pallidum antibody (TPAb)
8. Those who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, health products (except vitamin supplements) within 2 weeks before the first dose
9. Those who have a history of vaccination with live attenuated vaccine within 3 months before screening or a history of vaccination with inactivated vaccine within 1 month before screening
10. Those who have previously received dulaglutide or any other glucagon-like peptide-1 (GLP-1) analog
11. Those who donated blood or lost blood > or = 400 mL within 3 months before screening, or those who plan to donate blood
12. Those who smoked more than 5 cigarettes per day within 3 months before screening or who could not give up smoking during the period from signing the informed consent to the subjects leaving the group
13. Those who have a history of alcohol abuse, that is, drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine) , or those who have a positive alcohol breath test during the screening period
14. Those who have a history of drug abuse or poison use within 2 years before screening, or those who have a positive test results for urine drug abuse screening during the screening period
15. Participated in other clinical trials within 3 months before screening (subjects who are not randomized or not receiving treatment withdraw from the study before treatment, they can be enrolled in this study)
16. Acute illness or concomitant medication occurred from the time of signing the informed consent to the first administration
17. Those who have special requirements for diet and cannot obey the unified diet
18. Others judged by the investigator to be unsuitable to participate in this trial
19. Subjects who may not be able to complete this trial for other reasons

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Maximum (peak) plasma drug concentration(Cmax) | 0 hour (pre-dose,within 30mins) to 384 hours after administration
  Maximum (peak) plasma drug concentration
Area under the plasma concentration-time curve from time zero to ∞ (AUC0-∞) | 0 hour (pre-dose, within 30mins) to infinity
  The area under the plasma concentration curve from 0 to ∞

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | 0 hour (pre-dose,within 30mins) to 384 hours after administration
  The area under the plasma concentration curve from 0 to 384 h
Time to reach maximum plasma concentration following drug administration (Tmax) | 0 hour (pre-dose,within 30mins) to 384 hours after administration
  Time to maximum concentration
Elimination half-life (t1/2) | 0 hour (pre-dose,within 30mins) to 384 hours after administration
  Elimination half-life
Apparent total body clearance (CL/F) | 0 hour (pre-dose,within 30mins) to 384 hours after administration
  Apparent total body clearance
Apparent volume of distribution (Vd/F) | 0 hour (pre-dose,within 30mins) to 384 hours after administration
  Apparent volume of distribution
Elimination constants (λz) | 0 hour (pre-dose,within 30mins) to 384 hours after administration
  Elimination constants

CONTACTS AND LOCATIONS:
Overall Officials: Jie Hou, doctor, Principal Investigator — Peking University Care Luzhong Hospital; Hong Wang, bachelor, Principal Investigator — Peking University Care Luzhong Hospital
Locations (1):
- PKUCare Luzhong Hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] IDF (International Diabetes Federation) Diabetes Atlas, ninth edition, 2019.
- [Background] EMA. Trulicity® Risk Management Plan.2021.01.02.
- [Background] Geiser JS, Heathman MA, Cui X, Martin J, Loghin C, Chien JY, de la Pena A. Clinical Pharmacokinetics of Dulaglutide in Patients with Type 2 Diabetes: Analyses of Data from Clinical Trials. Clin Pharmacokinet. 2016 May;55(5):625-34. doi: 10.1007/s40262-015-0338-3. PMID 26507721
- [Background] FDA. Guidance for Industry - Clinical pharmacology data to support a demonstration of biosimilarity to a reference product. Dec. 2016.
- [Background] Barrington P, Chien JY, Tibaldi F, Showalter HD, Schneck K, Ellis B. LY2189265, a long-acting glucagon-like peptide-1 analogue, showed a dose-dependent effect on insulin secretion in healthy subjects. Diabetes Obes Metab. 2011 May;13(5):434-8. doi: 10.1111/j.1463-1326.2011.01365.x. Epub 2011 Jan 19. PMID 21251179
- [Background] Barrington P, Chien JY, Showalter HD, Schneck K, Cui S, Tibaldi F, Ellis B, Hardy TA. A 5-week study of the pharmacokinetics and pharmacodynamics of LY2189265, a novel, long-acting glucagon-like peptide-1 analogue, in patients with type 2 diabetes. Diabetes Obes Metab. 2011 May;13(5):426-33. doi: 10.1111/j.1463-1326.2011.01364.x. Epub 2011 Jan 19. PMID 21251178
- [Background] de la Pena A, Cui X, Geiser J, Loghin C. No Dose Adjustment is Recommended for Digoxin, Warfarin, Atorvastatin or a Combination Oral Contraceptive When Coadministered with Dulaglutide. Clin Pharmacokinet. 2017 Nov;56(11):1415-1427. doi: 10.1007/s40262-017-0531-7. PMID 28357715
- [Background] FDA (Food Drug Administration), Clinical Pharmacology Biopharmaceutics Review(s), 2014.
- [Background] EMA (European Medicines Agency), Public assessment report.2014
- [Derived] Gao X, Di Y, Lv Y, Luan Y, Xiong Y, Xu Y, Li Y, Guo L, Li X, Deng L, Zhuang Y, Hou J. A pharmacokinetic study comparing the biosimilar HEC14028 and Dulaglutide (Trulicity(R)) in healthy Chinese subjects. Clin Transl Sci. 2024 Apr;17(4):e13775. doi: 10.1111/cts.13775. PMID 38651744